CLINICAL TRIAL: NCT04727255
Title: Engaged and Resilient - a Preventive Resilience Intervention to Promote Psychological Well-being and Mental Health for Leaders in Organizations
Brief Title: Engaged and Resilient - a Preventive Intervention to Promote Psychological Well-being and Mental Health for Leaders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AU_IM
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-06

CONDITIONS: Stress, Psychological; Mental Health Issue
Keywords: Resilience; Positive mental health; Well-being
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized, controlled (two parallel groups)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will be implemented through a group-based delivery format involving internal educated resilience trainers. The Engaged and Resilient training program consists of twenty weekly, short-term sessions to build resilience skills in leaders.
  Interventions: Behavioral: Engaged and Resilient intervention
- Control (No Intervention): Participants in the (waitlist) control group will be exposed to their usual activities in the organization and will not perceive any interventions from the resilience curriculum. After the final data is collected, the control participant will be offered the opportunity to be trained by the internal trainers, educated in the research study.

INTERVENTIONS:
Behavioral: Engaged and Resilient intervention — Engaged and Resilient is a 3-phase program addressing the promotion of psychological resilience strategies for leaders.
  To implement resilience training as a strategic and ethical intervention in the organization, stakeholders from Management/HR will be involved in the final design of the training program based on local institutional data, and the baseline measure result. Local training sessions will be selected from a bag-log of resilience skills structured by three general resilience factors.
  To support ownership and internal sustainability, internal trainers will be educated on how to train the resilience skills in the program.
  The Engaged and Resilient program consists of 20 short-term sessions for leaders based on cognitive and positive psychology.
  Arms: Intervention

SUMMARY:
Leaders in organizations must handle organizational complexity and adversity as part of their position and profession. Work-related risk exposure is associated with perceived stress, low engagement, and mental health issues. However, not all leaders exposed to risk experience adverse outcomes, and one possible explanation might be their psychological ability to adapt to the organizational turbulence.

Engaged and Resilient is a research project for leaders in private and public organizations. The overall objective is to improve human health and performance, more specifically, to promote psychological and mental health by enhancing the resilience capacities to face adversity and adapt to the organizational environment. The Engaged and Resilient intervention is a flexible training program for leaders implemented as a 20-week program on-site (adjusted due to Covid-19).

DETAILED DESCRIPTION:
Research design:

The study involves program development, implementation, and evaluation of resilience training by a randomized controlled research design. The participant will be randomized to the intervention group to receive the resilience training program "Engaged and Resilient" or a wait-list control group to receive the resilience training conducted by internal educated trainers following the post-intervention measures.

Pre- and post measures include mental health, flourishing, perceived stress, resilience (two scales), and work-related performance (one-item). The training effects will be measured after each training session on a 4-point scale to create knowledge about the specific resilience promoting factors and the implementation process.

The intervention project will consist of an organizational supporting system and didactic component, including an internal trainer education for the Management/HR and more specific for the participants (leaders): Psychoeducation, psychological skill-building training, and ongoing homework exercises to support the implementation of resilience strategies within the organizational context.

Operational objectives:

* To develop a flexible (co-customized, co-implemented) resilience training program for leaders in organizations structured as thee general resilience factors with specific training sessions within each
* To implement a resilience intervention for leaders in public and private Danish organizational environments
* To demonstrate outcome effects on human health and performance. Primary in terms of mental health and well-being, and secondary in perceived stress, resilience, work-related performance, and sick-leave
* To provide evidence of specific resilience factors promoting positive mental health and well-being longitudinally (20 weeks)
* To create knowledge about the implementation and change process by ongoing participant evaluation of the specific training sessions

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Being a formal leader or having a specific leading role in a professional or functional area in the organization
* Accept the commitment to attendance in interventions groups and all sessions

Exclusion Criteria:

* Not willing and able to give informed consent
* Not willing to complete surveys at all time points

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in mental well-being | -1 month intervention (baseline), week 10, +1 month post intervention
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS-14) is a 14-item scale with 5 response categories.
Change in well-being (flourishing) | -1 month intervention (baseline), week 10, +1 month post intervention
  The Flourishing Scale is a 10-item scale with different (5,4 and 10) response categories.

SECONDARY OUTCOMES:
Change in perceived stress | -1 month intervention (baseline), week 10, +1 month post intervention
  The Perceived Stress Scale (PSS) is a 10-item scale with 5 response categories.
Change in work-related resilience | -1 month intervention (baseline), week 10, +1 month post intervention
  The resilience at work (RAW) Scale is a 20-item scale with 7 response categories.
Change in resilience | -1 month intervention (baseline), week 10, +1 month post intervention
  The CD-RISC 10 Scale is a 10-item scale with 5 response categories.
Job performance | -1 month intervention (baseline), week 10, +1 month post intervention
  The question on job performance (Pronk et al., 2004) has 10 response categories.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Henrik Knoop, Study Director — University of Aarhus
Locations (1):
- Aahus University, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No